CLINICAL TRIAL: NCT06816836
Title: Measuring Ultrasound Guided Skeletal Muscle Mass of Lower Extremity as a Predictor of Post-Operative Length of Stay in Exploratory Gynae-oncology Surgeries
Acronym: MUSLES
Status: Recruiting | Type: Observational
Sponsor: Tata Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/TMC/344/IRB66
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Gynecologic Cancer; Frailty; Sarcopenia
Keywords: Gynecologic Cancer; Post operative Stay; Frailty; Sarcopenia
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GC Patients, CCI Score 3+: All consecutive consenting Gynecological Cancer patients above 50 years of age undergoing open surgical intervention, with Charlson Co-morbidity Index score of 3 or more.
  Interventions: Procedure: Bed Side ultrasound guided muscle mass estimation of lower extremity

INTERVENTIONS:
Procedure: Bed Side ultrasound guided muscle mass estimation of lower extremity — Bed Side ultrasound guided muscle mass estimation of psoas major, rectus femoris, vastus intermedius and tibialis anterior.
  Other Names: Preoperative Charlson's comorbidity index scoring; Frailty by using Fried phenotype score; Markers of Sarcopenia from Abdominal pelvic CT scan

SUMMARY:
Increased incidence of Gynae-oncological cancer is observed specifically in women above 50 years of age. Sarcopenia (a progressive and generalized loss of skeletal muscle mass, quality, and strength) is considered a reliable indicator of frailty, a poor prognostic factor in these patients. Various frailty scores and measurement of psoas muscle mass are time consuming, can't be done in patients unable to walk and altered mental status. The investigators wanted to evaluate if bedside ultrasound guided skeletal muscle measurement, as a measure of sarcopenia, can be used to predict post operative length of stay.

DETAILED DESCRIPTION:
Gynae-oncological patients comprise a significant proportion of all new cancers and death related to cancer. Abrupt increase in the incidence of these cancer is observed specifically between women of 50-60 years of age. Therefore, it is important to evaluate the factors which influence postoperative outcomes in such patients. Sarcopenia, defined as a progressive and generalized loss of skeletal muscle mass, quality, and strength is considered a reliable indicator of frailty, a poor prognostic factor in cancer.

Usually, various frailty scores and measurement of psoas muscle mass with the abdominal pelvic CT scan are used as markers of sarcopenia. But these scores are time consuming, can't be done in patients unable to walk and altered mental status. Routine use of CT scan exposes the patient to radiation and may not be necessary.

The investigators wanted to evaluate if bedside ultrasound guided skeletal muscle measurement, as a measure of sarcopenia, can be used to predict adverse post operative outcomes in open gynae-oncology surgery in patients more than 50 years of age.

This will be a prospective observational cohort study. Total 320 patients will be recruited considering 1:1 ratio of sarcopenia vs non sarcopenia patients above the age of 50 years undergoing open gynae- oncology surgery.

The investigators will be collecting all relevant data other than skeletal muscle mass measurement (psoas major, rectus femoris, vastus intermedius and tibialis anterior) that can contribute to adverse post operative outcomes. In the preoperative period Charlson's comorbidity index, Serum albumin, creatinine and blood haemoglobin value, preoperative Functional status by 6-minute walk test, existing frailty by using Fried phenotype score and if patient has received neoadjuvant chemotherapy will be noted. Intraoperatively duration of surgery, Surgical complexity score, blood loss will be collected. In the post operative period,- length of hospital stay, Clavien Dindo score, Post operative morbidity score, 30 and 90 days readmission and 30 and 90 day mortality after discharge will be noted.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive consenting patients above 50 years of age, having a Charlson Comorbidity Index score of 3 or more, undergoing open surgeries for GCs.

Exclusion Criteria:

A. Refusal of consent B. Patients with psychiatric illnesses who are unable to follow instructions. C. Patients below the age of 50 years. D. Patients with known neuromuscular disorders. E. Patients in whom contrast-enhanced CT scan of the abdomen and pelvis is not done.

F. Previous major surgery of limbs (Amputation, Hip surgeries/ long bone surgeries)

Ages: 50 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above 50 years of age, with Charlson Comorbidity Index Score of 3 or more, presenting to the gynaecological oncology OPD with Gynacological Cancer to be treated with open surgery.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Prolonged length of hospital stay | 3 Years
  Length of hospital stay above 3rd Quartile at 9 days

SECONDARY OUTCOMES:
Incidence of severe morbidity as classified by the Clavien Dindo Score. | 3 years
  Incidence of severe morbidity as classified by the Clavien Dindo Score.
Type of morbidity as defined by the Post Operative Morbidity Survey. | 3 years
  Type of morbidity as defined by the Post Operative Morbidity Survey.
30-day and 90-day readmission | 3 years
  Readmission within 30 day/ 90 days from the day of discharge
30-day and 90-day mortality. | 3 years
  Mortality within 30 day/ 90 days from the day of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Medical Center, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: No